CLINICAL TRIAL: NCT02026063
Title: A Multicenter, Long-term Extension Study to Further Evaluate the Safety and Tolerability of Telotristat Etiprate (LX1606)
Brief Title: Telotristat Etiprate - Expanded Treatment for Patients With Carcinoid Syndrome Symptoms
Acronym: TELEPATH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LX1606.1-302-CS; LX1606.302 (Other: Lexicon Pharmaceuticals, Inc.); 2013-002596-18 (EudraCT Number)
Record Dates: First submitted 2013-12-31; First posted 2014-01-01 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-08

CONDITIONS: Carcinoid Syndrome
MeSH Terms: conditions — Serotonin Syndrome | interventions — telotristat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- 250 mg Telotristat Etiprate (Experimental): One telotristat etiprate (250 mg) tablet administered three times daily.
  Interventions: Drug: Telotristat etiprate
- 500 mg Telotristat Etiprate (Experimental): Two telotristat etiprate (250 mg) tablets administered three times daily.
  Interventions: Drug: Telotristat etiprate

INTERVENTIONS:
Drug: Telotristat etiprate — Telotristat etiprate tablet (250 mg)
  Other Names: LX1606

SUMMARY:
The primary objective of this study is to evaluate the long-term safety and tolerability of orally administered telotristat etiprate.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing participation in a Phase 2 [LX1606.1-202-CS (NCT00853047), LX1606.1-203-CS (NCT01104415)] or Phase 3 [LX1606.1-301-CS (NCT01677910), LX1606.1-303-CS (NCT02063659)] study
* Patients of childbearing potential must agree to use an adequate method of contraception (defined as having a failure rate of <1% per year) during the study and for 12 weeks after the Follow-up visit.
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Major protocol violations or tolerability concerns in a Phase 2 (eg, LX1606.1-202-CS, LX1606.1-203-CS) or Phase 3 (eg, LX1606.1-301-CS, LX1606.1-303-CS) study
* Positive pregnancy test
* Presence of any clinically significant findings at entry for medical history, laboratory values, or physical examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-01-14 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Lapuerta, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (40):
- United States (7):
  - Lexicon Investigational Site, Mobile, Alabama
  - Lexicon Investigational Site, Stanford, California
  - Lexicon Investigational Site, Iowa City, Iowa
  - Lexicon Investigational Site, Lexington, Kentucky
  - Lexicon Investigational Site, Boston, Massachusetts
  - Lexicon Investigational Site, New York, New York
  - Lexicon Investigational Site, Philadelphia, Pennsylvania
- Australia (3):
  - Lexicon Investigational Site, St Leonards, New South Wales
  - Lexicon Investigational Site, Herston, Queensland
  - Lexicon Investigational Site, East Melbourne, Victoria
- Belgium (3):
  - Lexicon Investigational Site, Edegem
  - Lexicon Investigational Site, Ghent
  - Lexicon Investigational Site, Yvoir
- Canada (2):
  - Lexicon Investgational Site, Calgary, Alberta
  - Lexicon Investigational Site, Halifax, Nova Scotia
- France (3):
  - Lexicon Investigational Site, Lille
  - Lexicon Investigational Site, Lyon
  - Lexicon Investigational Site, Villejuif
- Germany (5):
  - Lexicon Investigational Site, Bad Berka
  - Lexicon Investigational Site, Berlin
  - Lexicon Investigational Site, Essen
  - Lexicon Investigational Site, Hamburg
  - Lexicon Investigational Site, Marburg
- Lexicon Investigational Site, Jerusalem, Israel
- Italy (3):
  - Lexicon Investigational Site, Milan
  - Lexicon Investigational Site, Pisa
  - Lexicon Investigational Site, Torino
- Netherlands (3):
  - Lexicon Investigational Site, Amsterdam
  - Lexicon Investigational Site, Noord Holland
  - Lexicon Investigational Site, Noord-Brahant
- Spain (3):
  - Lexicon Investigational Site, Barcelona
  - Lexicon Investigational Site, Madrid
  - Lexicon Investigational Site, Seville
- Sweden (2):
  - Lexicon Investigational Site, Lund
  - Lexicon Investigational Site, Uppsala
- United Kingdom (5):
  - Lexicon Investigational Site, Coventry
  - Lexicon Investigational Site, Glasgow
  - Lexicon Investigational Site, London
  - Lexicon Investigational Site, Manchester
  - Lexicon Investigational Site, Newcastle upon Tyne

REFERENCES:
- [Derived] Horsch D, Anthony L, Gross DJ, Valle JW, Welin S, Benavent M, Caplin M, Pavel M, Bergsland E, Oberg K, Kassler-Taub KB, Binder P, Banks P, Lapuerta P, Kulke MH. Long-Term Treatment with Telotristat Ethyl in Patients with Carcinoid Syndrome Symptoms: Results from the TELEPATH Study. Neuroendocrinology. 2022;112(3):298-310. doi: 10.1159/000516958. Epub 2021 May 3. PMID 33940581

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants whose participation was ongoing in 1 of the following studies [LX1606.1-202-CS (NCT00853047), LX1606.1-203-CS (NCT01104415), LX1606.1-301-CS (NCT01677910), LX1606.1-303-CS (NCT02063659)] were eligible to enroll in this long-term safety study at the same dose received in the previous (parent) study.
Groups:
- Telotristat Etiprate 250 mg: Participants were treated with telotristat etiprate in a previous study for 9 to 46 months. Participants received one telotristat etiprate (250 mg) tablet three times daily (tid) up to an additional 228 weeks in this long-term extension study.
- Telotristat Etiprate 500 mg: Participants were treated with telotristat etiprate in a previous study for 9 to 46 months. Participants received two telotristat etiprate (250 mg) tablets tid up to an additional 204 weeks in this long-term extension study.
Period: Overall Study
Arm/Group | Telotristat Etiprate 250 mg | Telotristat Etiprate 500 mg
Started | 22 | 102
Completed | 13 | 53
Not Completed | 9 | 49
Not completed — Physician Decision | 0 | 10
Not completed — Noncompliance with Study Drug | 1 | 1
Not completed — Withdrawal of Consent | 1 | 6
Not completed — Adverse Event | 5 | 20
Not completed — Lack of Efficacy | 0 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Reason not Specified | 2 | 7

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received any fraction of a dose of telotristat etiprate during the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Telotristat Etiprate 250 mg | Telotristat Etiprate 500 mg | Total
Number analyzed (Participants) | 22 | 102 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (7.60) | 63.4 (10.33) | 63.6 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 41 | 55
  Male | 8 | 61 | 69
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 22 | 93 | 115
  Race: Black or African American | 0 | 2 | 2
  Race: American Indian or Alaska Native | 0 | 1 | 1
  Race: Other | 0 | 6 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 1 | 1
  Ethnicity: Not Hispanic or Latino | 22 | 100 | 122
  Ethnicity: Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 6 | 7
  Sweden | 0 | 8 | 8
  Netherlands | 1 | 8 | 9
  Belgium | 1 | 3 | 4
  United States | 3 | 28 | 31
  United Kingdom | 5 | 12 | 17
  Italy | 0 | 6 | 6
  Israel | 7 | 0 | 7
  France | 0 | 5 | 5
  Australia | 1 | 5 | 6
  Germany | 3 | 11 | 14
  Spain | 0 | 10 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE includes any noxious, pathological, or unintended change in anatomical, physiological, or metabolic functions as indicated by physical signs or symptoms occurring in any phase of the clinical study whether or not considered related to the study medication. A TEAE is an AE that occurs or worsens after receiving study drug.
Time Frame: First dose of study drug (Day 1) up to 15 days post last dose (approximately up to 236 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Telotristat Etiprate 250 mg | Telotristat Etiprate 500 mg
Number analyzed (Participants) | 22 | 102
Participants | 22 | 100

2. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) Score at Each Visit
Description: QLQ-C30 is a standardized 30-item scale to assess health-related quality of life composed of 5 functional scales (physical functioning [5 items], role functioning [2 items], emotional functioning [4 items], cognitive functioning [2 items], and social functioning [2 items]); 3 symptom scales (fatigue [3 items], nausea/vomiting [2 items], and pain [2 items]); a global health status (GHS) /quality of life (QOL) scale [2 items]; 6 single items (dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties). 28 questions answered:1 (not at all) to 4 (very much) and 2 questions on overall health/QOL answered:1 (poor) to 7 (excellent). All of the scales and single-item measures are transformed to a score:0 to 100. For functioning scales and global QOL higher scores indicate better functioning (a positive change from Baseline indicates improvement); for symptom scales higher scores indicate more severe symptoms (a negative change from Baseline indicates improvement).
Time Frame: Baseline, Weeks 24, 48, 72 and 84
Population: Per-Protocol (PP) population=participants who received telotristat etiprate;had no major protocol deviations that interfered with collection/interpretation of efficacy data. Number analyzed=participants with data at given time-point.Participants were combined for this outcome measure as they received dose adjustments per investigator's discretion.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Telotristat Etiprate (All Participants): Participants were treated with telotristat etiprate in a previous study for 9 to 46 months. Telotristat etiprate (250 or 500 mg) one or two tablets administered tid up to an additional 228 weeks (250 mg) or up to an additional 204 weeks (500 mg) in this long-term extension study.
Arm/Group | Telotristat Etiprate (All Participants)
Number analyzed (Participants) | 124
score on a scale
  GHS/QOL, Baseline: number analyzed (Participants) | 118
  GHS/QOL, Baseline | 60.664 (17.4627)
  GHS/QOL, Change at Week 24: number analyzed (Participants) | 102
  GHS/QOL, Change at Week 24 | -0.980 (17.9878)
  GHS/QOL, Change at Week 48: number analyzed (Participants) | 88
  GHS/QOL, Change at Week 48 | -4.261 (17.3239)
  GHS/QOL, Change at Week 72: number analyzed (Participants) | 77
  GHS/QOL, Change at Week 72 | -1.840 (17.0795)
  GHS/QOL, Change at Week 84: number analyzed (Participants) | 54
  GHS/QOL, Change at Week 84 | 0.309 (14.5660)
  Physical functioning, Baseline: number analyzed (Participants) | 120
  Physical functioning, Baseline | 79.958 (20.3109)
  Physical functioning, Change at Week 24: number analyzed (Participants) | 103
  Physical functioning, Change at Week 24 | -2.670 (13.6888)
  Physical functioning, Change at Week 48: number analyzed (Participants) | 90
  Physical functioning, Change at Week 48 | -2.667 (13.2129)
  Physical functioning, Change at Week 72: number analyzed (Participants) | 78
  Physical functioning, Change at Week 72 | -3.077 (14.8758)
  Physical functioning, Change at Week 84: number analyzed (Participants) | 55
  Physical functioning, Change at Week 84 | -1.939 (9.8275)
  Role functioning, Baseline: number analyzed (Participants) | 119
  Role functioning, Baseline | 73.810 (26.9766)
  Role functioning, Change at Week 24: number analyzed (Participants) | 102
  Role functioning, Change at Week 24 | -4.248 (23.9965)
  Role functioning, Change at Week 48: number analyzed (Participants) | 89
  Role functioning, Change at Week 48 | -5.431 (27.1518)
  Role functioning, Change at Week 72: number analyzed (Participants) | 77
  Role functioning, Change at Week 72 | -4.329 (23.9399)
  Role functioning, Change at Week 84: number analyzed (Participants) | 54
  Role functioning, Change at Week 84 | -1.543 (21.5414)
  Emotional functioning, Baseline: number analyzed (Participants) | 118
  Emotional functioning, Baseline | 75.683 (21.6630)
  Emotional functioning, Change at Week 24: number analyzed (Participants) | 102
  Emotional functioning, Change at Week 24 | -1.552 (17.5010)
  Emotional functioning, Change at Week 48: number analyzed (Participants) | 88
  Emotional functioning, Change at Week 48 | -0.852 (17.5549)
  Emotional functioning, Change at Week 72: number analyzed (Participants) | 77
  Emotional functioning, Change at Week 72 | -1.623 (19.7313)
  Emotional functioning, Change at Week 84: number analyzed (Participants) | 54
  Emotional functioning, Change at Week 84 | 3.858 (14.3621)
  Cognitive functioning, Baseline: number analyzed (Participants) | 118
  Cognitive functioning, Baseline | 78.955 (21.7283)
  Cognitive functioning, Change at Week 24: number analyzed (Participants) | 102
  Cognitive functioning, Change at Week 24 | 0.000 (18.1668)
  Cognitive functioning, Change at Week 48: number analyzed (Participants) | 88
  Cognitive functioning, Change at Week 48 | -1.515 (16.8830)
  Cognitive functioning, Change at Week 72: number analyzed (Participants) | 77
  Cognitive functioning, Change at Week 72 | -1.299 (22.2568)
  Cognitive functioning, Change at Week 84: number analyzed (Participants) | 54
  Cognitive functioning, Change at Week 84 | 3.086 (18.0478)
  Social functioning, Baseline: number analyzed (Participants) | 118
  Social functioning, Baseline | 74.011 (24.1220)
  Social functioning, Change at Week 24: number analyzed (Participants) | 102
  Social functioning, Change at Week 24 | -1.797 (21.2258)
  Social functioning, Change at Week 48: number analyzed (Participants) | 88
  Social functioning, Change at Week 48 | -4.167 (24.5327)
  Social functioning, Change at Week 72: number analyzed (Participants) | 77
  Social functioning, Change at Week 72 | -1.732 (26.0151)
  Social functioning, Change at Week 84: number analyzed (Participants) | 54
  Social functioning, Change at Week 84 | -0.617 (20.7215)
  Fatigue, Baseline: number analyzed (Participants) | 120
  Fatigue, Baseline | 33.981 (24.7530)
  Fatigue, Change at Week 24: number analyzed (Participants) | 103
  Fatigue, Change at Week 24 | 4.800 (21.3903)
  Fatigue, Change at Week 48: number analyzed (Participants) | 90
  Fatigue, Change at Week 48 | 7.284 (20.9473)
  Fatigue, Change at Week 72: number analyzed (Participants) | 78
  Fatigue, Change at Week 72 | 6.054 (19.3320)
  Fatigue, Change at Week 84: number analyzed (Participants) | 55
  Fatigue, Change at Week 84 | 4.444 (17.8394)
  Nausea and vomiting, Baseline: number analyzed (Participants) | 119
  Nausea and vomiting, Baseline | 9.104 (13.3312)
  Nausea and vomiting, Change at Week 24: number analyzed (Participants) | 103
  Nausea and vomiting, Change at Week 24 | 1.618 (15.0371)
  Nausea and vomiting, Change at Week 48: number analyzed (Participants) | 90
  Nausea and vomiting, Change at Week 48 | 0.556 (14.8757)
  Nausea and vomiting, Change at Week 72: number analyzed (Participants) | 78
  Nausea and vomiting, Change at Week 72 | 2.137 (20.3432)
  Nausea and vomiting, Change at Week 84: number analyzed (Participants) | 55
  Nausea and vomiting, Change at Week 84 | -1.212 (15.3339)
  Pain, Baseline: number analyzed (Participants) | 120
  Pain, Baseline | 26.528 (25.0579)
  Pain, Change at Week 24: number analyzed (Participants) | 103
  Pain, Change at Week 24 | 3.722 (21.8845)
  Pain, Change at Week 48: number analyzed (Participants) | 90
  Pain, Change at Week 48 | 6.481 (22.9930)
  Pain, Change at Week 72: number analyzed (Participants) | 78
  Pain, Change at Week 72 | 1.709 (26.5351)
  Pain, Change at Week 84: number analyzed (Participants) | 55
  Pain, Change at Week 84 | -4.848 (22.3774)
  Dyspnea, Baseline: number analyzed (Participants) | 120
  Dyspnea, Baseline | 18.611 (24.7474)
  Dyspnea, Change at Week 24: number analyzed (Participants) | 103
  Dyspnea, Change at Week 24 | 1.294 (19.7602)
  Dyspnea, Change at Week 48: number analyzed (Participants) | 89
  Dyspnea, Change at Week 48 | 5.618 (22.0399)
  Dyspnea, Change at Week 72: number analyzed (Participants) | 78
  Dyspnea, Change at Week 72 | 2.564 (21.3331)
  Dyspnea, Change at Week 84: number analyzed (Participants) | 55
  Dyspnea, Change at Week 84 | 6.667 (16.2288)
  Insomnia, Baseline: number analyzed (Participants) | 120
  Insomnia, Baseline | 26.389 (28.6307)
  Insomnia, Change at Week 24: number analyzed (Participants) | 103
  Insomnia, Change at Week 24 | 3.560 (26.3679)
  Insomnia, Change at Week 48: number analyzed (Participants) | 90
  Insomnia, Change at Week 48 | 3.704 (27.1144)
  Insomnia, Change at Week 72: number analyzed (Participants) | 78
  Insomnia, Change at Week 72 | 2.564 (24.4827)
  Insomnia, Change at Week 84: number analyzed (Participants) | 55
  Insomnia, Change at Week 84 | 0.000 (21.2762)
  Appetite loss, Baseline: number analyzed (Participants) | 119
  Appetite loss, Baseline | 13.165 (21.3563)
  Appetite loss, Change at Week 24: number analyzed (Participants) | 102
  Appetite loss, Change at Week 24 | 3.595 (26.0772)
  Appetite loss, Change at Week 48: number analyzed (Participants) | 89
  Appetite loss, Change at Week 48 | 3.745 (21.5780)
  Appetite loss, Change at Week 72: number analyzed (Participants) | 78
  Appetite loss, Change at Week 72 | 10.256 (27.5543)
  Appetite loss, Change at Week 84: number analyzed (Participants) | 55
  Appetite loss, Change at Week 84 | 4.848 (22.6061)
  Constipation, Baseline: number analyzed (Participants) | 118
  Constipation, Baseline | 7.345 (16.3854)
  Constipation, Change at Week 24: number analyzed (Participants) | 102
  Constipation, Change at Week 24 | 3.595 (18.7079)
  Constipation, Change at Week 48: number analyzed (Participants) | 88
  Constipation, Change at Week 48 | 0.379 (17.8645)
  Constipation, Change at Week 72: number analyzed (Participants) | 77
  Constipation, Change at Week 72 | 4.762 (20.7423)
  Constipation, Change at Week 84: number analyzed (Participants) | 54
  Constipation, Change at Week 84 | 3.086 (19.7134)
  Diarrhea, Baseline: number analyzed (Participants) | 118
  Diarrhea, Baseline | 42.090 (33.3128)
  Diarrhea, Change at Week 24: number analyzed (Participants) | 102
  Diarrhea, Change at Week 24 | 1.961 (29.9701)
  Diarrhea, Change at Week 48: number analyzed (Participants) | 88
  Diarrhea, Change at Week 48 | 5.682 (34.7300)
  Diarrhea, Change at Week 72: number analyzed (Participants) | 76
  Diarrhea, Change at Week 72 | 3.947 (32.1879)
  Diarrhea, Change at Week 84: number analyzed (Participants) | 53
  Diarrhea, Change at Week 84 | 0.000 (31.3513)
  Financial difficulties, Baseline: number analyzed (Participants) | 118
  Financial difficulties, Baseline | 18.079 (28.1240)
  Financial difficulties, Change at Week 24: number analyzed (Participants) | 102
  Financial difficulties, Change at Week 24 | -0.327 (15.9034)
  Financial difficulties, Change at Week 48: number analyzed (Participants) | 87
  Financial difficulties, Change at Week 48 | 1.533 (19.6270)
  Financial difficulties, Change at Week 72: number analyzed (Participants) | 77
  Financial difficulties, Change at Week 72 | 0.433 (25.0692)
  Financial difficulties, Change at Week 84: number analyzed (Participants) | 54
  Financial difficulties, Change at Week 84 | -1.235 (19.3857)

3. Secondary Outcome: Change From Baseline in Gastrointestinal Symptoms of Carcinoid Neuroendocrine Tumors (GI.NET21) Score at Each Visit
Description: GI.NET21 is a standardized 21-item scale composed of both multi-item scales and single-item measures that include 5 functional scales (gastrointestinal (GI) [5 items], endocrine [3 items], treatment-related [3 items], social functioning [3 items], and disease-related worries scale [DRWS] [3 items]) and 4 single items (muscle and bone pain symptom (BPS), sexual functioning, communication function (CF), body image and information about the disease). Each item is scored from 1 (not at all) to 4 (very much). All of the scales and single-item measures are transformed to a score of 0 to 100. For functioning scales higher scores indicate better functioning (a positive change from Baseline indicates improvement); for symptom scales higher scores indicate more severe symptoms (a negative change from Baseline indicates improvement).
Time Frame: Baseline, Weeks 24, 48, 72 and 84
Population: PP population included the participants who received telotristat etiprate; had no major protocol deviations that interfered with collection/interpretation of efficacy data. Number analyzed=participants with data at given time-point. Participants were combined for this outcome measure as they received dose adjustments per investigator's discretion.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telotristat Etiprate (All Participants)
Number analyzed (Participants) | 124
score on a scale
  Endocrine scale, Baseline: number analyzed (Participants) | 120
  Endocrine scale, Baseline | 25.000 (20.6367)
  Endocrine scale, Change at Week 24: number analyzed (Participants) | 103
  Endocrine scale, Change at Week 24 | 1.726 (15.8483)
  Endocrine scale, Change at Week 48: number analyzed (Participants) | 90
  Endocrine scale, Change at Week 48 | 1.111 (17.0717)
  Endocrine scale, Change at Week 72: number analyzed (Participants) | 78
  Endocrine scale, Change at Week 72 | 1.425 (19.8082)
  Endocrine scale, Change at Week 84: number analyzed (Participants) | 54
  Endocrine scale, Change at Week 84 | 4.938 (21.2213)
  GI symptoms scale, Baseline: number analyzed (Participants) | 120
  GI symptoms scale, Baseline | 25.014 (17.9343)
  GI symptoms scale, Change at Week 24: number analyzed (Participants) | 103
  GI symptoms scale, Change at Week 24 | 3.576 (14.9243)
  GI symptoms scale, Change at Week 48: number analyzed (Participants) | 90
  GI symptoms scale, Change at Week 48 | 3.759 (16.7890)
  GI symptoms scale, Change at Week 72: number analyzed (Participants) | 78
  GI symptoms scale, Change at Week 72 | 1.581 (19.0823)
  GI symptoms scale, Change at Week 84: number analyzed (Participants) | 54
  GI symptoms scale, Change at Week 84 | -0.278 (17.3137)
  Treatment scale, Baseline: number analyzed (Participants) | 101
  Treatment scale, Baseline | 10.176 (14.6370)
  Treatment scale, Change at Week 24: number analyzed (Participants) | 80
  Treatment scale, Change at Week 24 | -0.486 (13.7849)
  Treatment scale, Change at Week 48: number analyzed (Participants) | 66
  Treatment scale, Change at Week 48 | 1.684 (14.0873)
  Treatment scale, Change at Week 72: number analyzed (Participants) | 58
  Treatment scale, Change at Week 72 | 0.575 (18.8668)
  Treatment scale, Change at Week 84: number analyzed (Participants) | 35
  Treatment scale, Change at Week 84 | 2.063 (20.4384)
  Social function scale, Baseline: number analyzed (Participants) | 120
  Social function scale, Baseline | 32.037 (22.8748)
  Social function scale, Change at Week 24: number analyzed (Participants) | 103
  Social function scale, Change at Week 24 | 3.128 (16.4229)
  Social function scale, Change at Week 48: number analyzed (Participants) | 90
  Social function scale, Change at Week 48 | 2.160 (22.4658)
  Social function scale, Change at Week 72: number analyzed (Participants) | 77
  Social function scale, Change at Week 72 | 1.587 (21.3052)
  Social function scale, Change at Week 84: number analyzed (Participants) | 54
  Social function scale, Change at Week 84 | 0.000 (18.4415)
  DRWS, Baseline: number analyzed (Participants) | 120
  DRWS, Baseline | 36.713 (26.9224)
  DRWS, Change at Week 24: number analyzed (Participants) | 103
  DRWS, Change at Week 24 | 1.456 (20.4932)
  DRWS, Change at Week 48: number analyzed (Participants) | 90
  DRWS, Change at Week 48 | -1.049 (22.5767)
  DRWS, Change at Week 72: number analyzed (Participants) | 77
  DRWS, Change at Week 72 | -0.289 (26.5962)
  DRWS, Change at Week 84: number analyzed (Participants) | 54
  DRWS, Change at Week 84 | -3.601 (22.4868)
  Muscle and BPS, Baseline: number analyzed (Participants) | 120
  Muscle and BPS, Baseline | 30.833 (27.7250)
  Muscle and BPS, Change at Week 24: number analyzed (Participants) | 102
  Muscle and BPS, Change at Week 24 | -3.268 (21.7546)
  Muscle and BPS, Change at Week 48: number analyzed (Participants) | 90
  Muscle and BPS, Change at Week 48 | 7.407 (31.9088)
  Muscle and BPS, Change at Week 72: number analyzed (Participants) | 76
  Muscle and BPS, Change at Week 72 | -1.316 (25.2048)
  Muscle and BPS, Change at Week 84: number analyzed (Participants) | 54
  Muscle and BPS, Change at Week 84 | 2.469 (24.9543)
  Sexual function, Baseline: number analyzed (Participants) | 91
  Sexual function, Baseline | 30.769 (36.5928)
  Sexual function, Change at Week 24: number analyzed (Participants) | 62
  Sexual function, Change at Week 24 | 2.151 (29.4893)
  Sexual function, Change at Week 48: number analyzed (Participants) | 58
  Sexual function, Change at Week 48 | -2.299 (24.0711)
  Sexual function, Change at Week 72: number analyzed (Participants) | 51
  Sexual function, Change at Week 72 | -3.922 (24.6280)
  Sexual function, Change at Week 84: number analyzed (Participants) | 36
  Sexual function, Change at Week 84 | -1.852 (19.4274)
  Information and CF, Baseline: number analyzed (Participants) | 120
  Information and CF, Baseline | 2.500 (9.8186)
  Information and CF, Change at Week 24: number analyzed (Participants) | 103
  Information and CF, Change at Week 24 | 3.236 (17.1591)
  Information and CF, Change at Week 48: number analyzed (Participants) | 90
  Information and CF, Change at Week 48 | 0.741 (13.1995)
  Information and CF, Change at Week 72: number analyzed (Participants) | 77
  Information and CF, Change at Week 72 | 1.299 (13.7241)
  Information and CF, Change at Week 84: number analyzed (Participants) | 54
  Information and CF, Change at Week 84 | 5.556 (25.6978)
  Body image, Baseline: number analyzed (Participants) | 119
  Body image, Baseline | 11.765 (21.5187)
  Body image, Change at Week 24: number analyzed (Participants) | 100
  Body image, Change at Week 24 | 6.333 (24.4789)
  Body image, Change at Week 48: number analyzed (Participants) | 89
  Body image, Change at Week 48 | 5.618 (23.1573)
  Body image, Change at Week 72: number analyzed (Participants) | 76
  Body image, Change at Week 72 | 6.579 (28.8134)
  Body image, Change at Week 84: number analyzed (Participants) | 53
  Body image, Change at Week 84 | 3.774 (27.4721)

4. Secondary Outcome: Percentage of Participants With Adequate Relief as Per Subjective Global Assessment Question
Description: Participants were asked to respond to the following question: "In the past 7 days, have you had adequate relief of your carcinoid syndrome bowel complaints such as diarrhea, urgent need to have a bowel movement, abdominal pain, or discomfort? The percentage of participants reporting adequate relief (answered Yes) were reported.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72 and 84
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Telotristat Etiprate (All Participants)
Number analyzed (Participants) | 124
percentage of participants
  Baseline: number analyzed (Participants) | 99
  Baseline | 61.6
  Week 12: number analyzed (Participants) | 106
  Week 12 | 64.2
  Week 24: number analyzed (Participants) | 104
  Week 24 | 52.9
  Week 36: number analyzed (Participants) | 95
  Week 36 | 57.9
  Week 48: number analyzed (Participants) | 95
  Week 48 | 61.1
  Week 60: number analyzed (Participants) | 89
  Week 60 | 55.1
  Week 72: number analyzed (Participants) | 77
  Week 72 | 58.4
  Week 84: number analyzed (Participants) | 55
  Week 84 | 67.3

5. Secondary Outcome: Change From Baseline in Subjective Global Assessment of Carcinoid Syndrome Symptoms on 11-Point Numeric Scale at Each Visit
Description: Participants were asked the following question to assess global symptoms associated with carcinoid syndrome (CS) on an 11-point scale: "Rate the severity of your overall carcinoid symptoms over the past 7 days on a scale from 0 to 10, where 0=no symptoms and 10=worst symptoms ever experienced. A negative change from baseline indicated improvement.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72 and 84
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telotristat Etiprate (All Participants)
Number analyzed (Participants) | 124
score on a scale
  Baseline: number analyzed (Participants) | 92
  Baseline | 3.022 (1.9214)
  Change at Week 12: number analyzed (Participants) | 86
  Change at Week 12 | 0.558 (2.4428)
  Change at Week 24: number analyzed (Participants) | 78
  Change at Week 24 | 0.654 (2.2553)
  Change at Week 36: number analyzed (Participants) | 73
  Change at Week 36 | 0.630 (2.2944)
  Change at Week 48: number analyzed (Participants) | 71
  Change at Week 48 | 1.056 (2.5684)
  Change at Week 60: number analyzed (Participants) | 66
  Change at Week 60 | 0.576 (1.9773)
  Change at Week 72: number analyzed (Participants) | 60
  Change at Week 72 | 0.483 (2.2661)
  Change at Week 84: number analyzed (Participants) | 45
  Change at Week 84 | 0.644 (2.2172)

ADVERSE EVENTS:
Time Frame: First dose of study drug (Day 1) up to 15 days post last dose (approximately up to 236 weeks)
Description: Safety population included all participants who received any fraction of a dose of telotristat etiprate during the study.
Arm/Group | Telotristat Etiprate 250 mg | Telotristat Etiprate 500 mg
All-Cause Mortality (participants affected / at risk) | 2/22 | 18/102
Serious Adverse Events (participants affected / at risk) | 12/22 | 54/102
Other Adverse Events (participants affected / at risk) | 22/22 | 100/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telotristat Etiprate 250 mg (N=22) | Telotristat Etiprate 500 mg (N=102)
Embolism (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Radiotherapy (Surgical and medical procedures) | 0 | 2
Ileocolectomy (Surgical and medical procedures) | 0 | 1
Investigation (Investigations) | 1 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to testicle (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1
Disease progression (General disorders) | 2 | 11
General physical health deterioration (General disorders) | 0 | 3
Death (General disorders) | 0 | 2
Complication of device insertion (General disorders) | 0 | 1
Device failure (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
General physical condition abnormal (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Laparoscopy (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 2
Haemorrhagic stroke (Nervous system disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 6
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Subileus (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 2
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basedow's disease (Endocrine disorders) | 1 | 0
Carcinoid crisis (Endocrine disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 3
Sepsis (Infections and infestations) | 1 | 2
Abdominal wall abscess (Infections and infestations) | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 1
Perihepatic abscess (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telotristat Etiprate 250 mg (N=22) | Telotristat Etiprate 500 mg (N=102)
Flushing (Vascular disorders) | 4 | 13
Hypertension (Vascular disorders) | 1 | 13
Radiotherapy (Surgical and medical procedures) | 2 | 2
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Fatigue (General disorders) | 4 | 28
Pyrexia (General disorders) | 1 | 20
Disease progression (General disorders) | 2 | 16
Oedema peripheral (General disorders) | 1 | 17
Asthenia (General disorders) | 0 | 15
Chest discomfort (General disorders) | 2 | 2
Depression (Psychiatric disorders) | 2 | 11
Depressed mood (Psychiatric disorders) | 0 | 9
Insomnia (Psychiatric disorders) | 1 | 8
Weight decreased (Investigations) | 1 | 15
Gamma-glutamyltransferase increased (Investigations) | 3 | 3
Investigation (Investigations) | 3 | 3
Blood glucose increased (Investigations) | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 10
Dizziness (Nervous system disorders) | 1 | 10
Headache (Nervous system disorders) | 1 | 10
Syncope (Nervous system disorders) | 1 | 10
Diarrhoea (Gastrointestinal disorders) | 9 | 35
Nausea (Gastrointestinal disorders) | 5 | 36
Abdominal pain (Gastrointestinal disorders) | 3 | 37
Constipation (Gastrointestinal disorders) | 3 | 22
Vomiting (Gastrointestinal disorders) | 1 | 24
Abdominal pain upper (Gastrointestinal disorders) | 2 | 13
Flatulence (Gastrointestinal disorders) | 1 | 7
Abdominal distension (Gastrointestinal disorders) | 0 | 6
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 6
Glossodynia (Gastrointestinal disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 8
Rash (Skin and subcutaneous tissue disorders) | 0 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 15
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 8
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 3 | 13
Dehydration (Metabolism and nutrition disorders) | 0 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 6
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 6
Nasopharyngitis (Infections and infestations) | 2 | 9
Urinary tract infection (Infections and infestations) | 2 | 9
Influenza (Infections and infestations) | 2 | 8
Upper respiratory tract infection (Infections and infestations) | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any confidential information, proprietary information, or patentable subject matter.

DOCUMENTS (2):
  • Study Protocol (2015-11-02): https://cdn.clinicaltrials.gov/large-docs/63/NCT02026063/Prot_000.pdf
  • Statistical Analysis Plan (2014-11-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT02026063/SAP_001.pdf